CLINICAL TRIAL: NCT02441309
Title: A Mechanistic Study Of Mifamurtide (MTP-PE) In Patients With Metastatic And/Or Recurrent Osteosarcoma
Brief Title: A Eurosarc Study of Mifamurtide in Advanced Osteosarcoma (MEMOS)
Acronym: MEMOS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failed to recruit sufficient numbers of patients in the funded period
Sponsor: University of Oxford (Other)
Collaborators: Millennium: The Takeda Oncology Company (Industry); National Institute for Health Research, United Kingdom (Other Government); Oxford University Hospitals NHS Trust (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_039
Record Dates: First submitted 2015-03-16; First posted 2015-05-12 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-03

CONDITIONS: Osteosarcoma
Keywords: Metastatic and/or Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — mifamurtide; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A. Mifamurtide only (Experimental): Treatment Weeks 1-6 (post 1st biopsy/resection):
  Mifamurtide 2mg/m2, IV infusion, twice/week, with each infusion given at least 3 days apart, for 6 weeks.
  Treatment Weeks 7-12 (post 2nd biopsy/resection):
  Mifamurtide 2mg/m2, IV infusion, twice/week, with each infusion given at least 3 days apart, for 6 weeks.
  Treatment Weeks 13-36:
  Mifamurtide 2mg/m2, IV infusion, once/week.
  Interventions: Drug: Mifamurtide
- B. Ifosfamide (Followed by Mifamurtide) (Experimental): Treatment Weeks 1-6: Day 1 of 21: Ifosfamide 12-15g/m2 IV infused over 4-5 days as per local practice. Repeated every 21 days for 2 cycles (3 weeks=1 cycle).
  Treatment Weeks 7-12 (post 2nd biopsy/resection): Day 1 of 21: Ifosfamide 12-15g/m2 IV infused over 4-5 days once every 21 days for two cycles (3 weeks=1 cycle). Ifosfamide administered as per local practice, including concurrent dosing with mesna. Plus mifamurtide 2mg/m2, IV infusion, twice/week. Ifosfamide infusion started 24 hours prior to mifamurtide. Mifamurtide given on day 2 and either day 5 or day 6.
  Treatment Weeks 13-18: Mifamurtide 2mg/m2, IV infusion, twice/week. Treatment Weeks 19-42: Mifamurtide 2mg/m2, IV infusion, once/week.
  Interventions: Drug: Mifamurtide; Drug: Ifosfamide
- C. Ifosfamide + Mifamurtide (Experimental): Treatment Weeks 1-6:
  Day 1 of 21: Ifosfamide 12-15g/m2 IV infusion over 4-5 days once every 21 days for two cycles (3 weeks=1 cycle).
  Plus Mifamurtide 2mg/m2, IV infusion, twice per week, each given at least 3 days apart, for 6 weeks.
  Ifosfamide infusion started 24 hours prior to mifamurtide. Mifamurtide given on day 2 and either day 5 or day 6.
  Treatment Weeks 7-12 (post 2nd biopsy/resection):
  Day 1 of 21: Ifosfamide 12-15g/m2 IV infusion over 4-5 days once every 21 days for two cycles (3 weeks = 1 cycle).
  Plus Mifamurtide 2mg/m2, IV infusion, twice per week, given at least 3 days apart, for 6 weeks. Ifosfamide infusion started 24 hours prior to mifamurtide. Mifamurtide given on day 2 and either day 5 or day 6.
  Treatment Weeks 13-36: Mifamurtide 2mg/m2, IV infusion, once/week.
  Interventions: Drug: Mifamurtide; Drug: Ifosfamide

INTERVENTIONS:
Drug: Mifamurtide
Drug: Ifosfamide
  Arms: B. Ifosfamide (Followed by Mifamurtide); C. Ifosfamide + Mifamurtide

SUMMARY:
This is a Bayesian designed multi-arm, multi-centre, open label phase II study. The target sample size of 40 patients will be recruited from up to 8 EU countries, but this may be revised in light of the interim analysis. Patients with relapsed or metastatic osteosarcoma will be divided into three treatment groups. They will all either have surgery or a biopsy before and after six weeks exposure to either Mifamurtide alone, Ifosfamide alone, or Mifamurtide combined with Ifosfamide. They will then receive further treatment to a maximum of 42 or 36 weeks in total (depending on Arm), with all patients being able to receive 36 weeks of Mifamurtide treatment.

DETAILED DESCRIPTION:
Osteosarcoma (OS) is the most common primary tumour arising from bones. There is currently no approved treatment other than surgery for metastatic or recurrent osteosarcoma refractory to chemotherapy. Patients deemed unresectable normally receive chemotherapy prior to attempted resection. The addition of chemotherapy to surgery for metastatic or recurrent osteosarcoma may improve response rates. MEPACT (Mifamurtide, MTP-PE) is licensed for use in the adjuvant osteosarcoma setting; indicated in children, adolescents and young adults for the treatment of high-grade resectable non-metastatic osteosarcoma after macroscopically complete surgical resection. It is used in combination with post-operative multi-agent chemotherapy. This is a Bayesian designed multi-arm, multi-centre open-label phase II study in patients with metastatic and/or recurrent osteosarcoma, which will investigate why some patients with osteosarcoma may respond better than others to mifamurtide given alone or in combination with ifosfamide. Patients with relapsed or metastatic osteosarcoma will be divided into three treatment groups (Arms). Depending on their current disease status, patients may be either Registered to Arm A (resectable group), to receive Mifamurtide alone; or Randomised to Arm B/C (non-resectable group), to receive mifamurtide in combination with ifosfamide. Arm A - Mifamurtide alone; Arm B - Ifosfamide alone for 6 weeks then Ifosfamide + mifamurtide for 6 weeks, then mifamurtide alone for 30 weeks; Arm C - Ifosfamide + mifamurtide for 12 weeks then mifamurtide alone for 24 weeks. All participants will receive 36 weeks or more of mifamurtide. Biopsies (or resected tumour samples) will be obtained before and after 6 weeks of therapy interval in order to determine the pharmacodynamic endpoints. The target sample size is 40 patients. An interim analysis will be performed for the primary efficacy endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed osteosarcoma (first, second, third or any relapse, patient has recovered from chemotherapy and any other investigational drug/agent treatment, radiotherapy or surgical procedure).
2. Histological confirmed diagnosis of osteosarcoma at original presentation.
3. Tumour at biopsy accessible or resectable site.
4. Progressive disease documented by imaging within 3 months of entry into the trial.
5. At least one measurable lesion on CT scan (RECIST) performed in past 21 days prior to trial entry.
6. Male or female, age ≥ 16 years to 65 (or ≥18 based on institutional practice for Teenage and Young Adult Cancer patients).
7. Life expectancy of at least 3 months.
8. WHO performance score of 0 - 2.
9. The patient is willing and able to comply with the protocol and scheduled follow-up visits and examinations.
10. Written (signed and dated) informed consent.
11. Cardiac shortening fraction ≥ 28% or ejection fraction ≥ 45%
12. Renal function is adequate for ifosfamide treatment (GFR as per table below, other renal function screening tests as per local practice)
13. Haematological and biochemical indices within the ranges shown below:

Lab Test Value required

* Haemoglobin (Hb) ≥ 9 g/dL (Previous transfusion is allowed)
* Absolute neutrophil count (ANC) >=1.0 x 10*9/L without growth factor support
* Platelet count > 80.x 10*9/L (Previous transfusion is allowed)
* Total bilirubin <1.5 times the upper limit of normal (ULN) for age (except for Gilbert's syndrome patients)
* Serum alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) <2.5 × ULN for age, <2.5 × ULN for age
* Serum creatinine Normal range for age
* Glomerular filtration rate (GFR) (calculated as 51Cr-EDTA/99mTc-DTPA clearance) >40ml/min if deemed resectable (for Arm A), >60ml/min if not deemed resectable (for Arm B or C)

Exclusion Criteria:

1. Pregnant or breast-feeding woman. Men or women of childbearing potential unless effective methods of contraception are used during study treatment and for at least 7 days after the last mifamurtide dose (see section 5.1 Informed consent - Contraceptive/ Pregnancy counselling).
2. Previous treatment with mifamurtide or a mifamurtide-like drug* in a clinical trial setting for the treatment of metastatic and/or recurrent osteosarcoma in the six months prior to registration.
3. Contraindications to lung biopsies.
4. Hypersensitivity to ifosfamide or any component of the formulation.
5. Previously diagnosed brain metastases.
6. Significant active cardiac disease including: uncontrolled high blood pressure (no greater than 2 standard deviations above the mean for age for systolic blood pressure (SBP) and diastolic blood pressure (DBP), unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, or serious cardiac arrhythmias and with a history of pericarditis and myocarditis
7. Treatment with any other investigational agent, or participation in another interventional clinical trial within 21 days prior to enrolment.
8. Major surgery within 21 days prior to first study biopsy
9. Currently taking high-dose non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroid treatment
10. Concurrent use of ciclosporin or other calcineurin inhibitors.
11. Any psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
12. Any other active malignancy, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and non-melanoma skin lesions.
13. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.

    * mifamurtide-like drugs include GCSF, GMCSF, interferon and other macrophage activating molecules.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bass Hassan, BMBCh FRCP, Principal Investigator — University of Oxford
Locations (8):
- Pediatric Hematology and Oncology, University Hospital Münster, Münster, Germany
- Istituti Ortopedici Rizzoli, Bologna, Emilia-Romagna, Italy
- Department of Clinical Oncology, Leiden University Medical Center, Leiden, Postzone K1-P, Netherlands
- Radium Hospital, Oslo University, Oslo, Norway
- United Kingdom (4):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University College London Hospitals NHS Foundation Trust, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundations Trust, Oxford

RESULTS

PARTICIPANT FLOW:
Groups:
- A. Mifamurtide Only: Patients receive Mifamurtide only.
  Treatment Weeks 1-6 (post 1st biopsy/resection):
  Mifamurtide 2mg/m2, IV infusion, twice/week, with each infusion given at least 3 days apart, for 6 weeks.
  Treatment Weeks 7-12 (post 2nd biopsy/resection):
  Mifamurtide 2mg/m2, IV infusion, twice/week, with each infusion given at least 3 days apart, for 6 weeks.
  Treatment Weeks 13-36:
  Mifamurtide 2mg/m2, IV infusion, once/week.
  Mifamurtide
- B. Ifosfamide (Followed by Mifamurtide): Patients receive Ifosfamide alone initially, followed by ifosfamide plus mifamurtide, then mifamurtide alone.
  Treatment Weeks 1-6: Day 1 of 21: Ifosfamide 12-15g/m2 IV infused over 4-5 days as per local practice. Repeated every 21 days for 2 cycles (3 weeks=1 cycle).
  Treatment Weeks 7-12 (post 2nd biopsy/resection): Day 1 of 21: Ifosfamide 12-15g/m2 IV infused over 4-5 days once every 21 days for two cycles (3 weeks=1 cycle). Ifosfamide administered as per local practice, including concurrent dosing with mesna. Plus mifamurtide 2mg/m2, IV infusion, twice/week. Ifosfamide infusion must be started 24 hours prior to mifamurtide. Mifamurtide should be given on day 2 and either day 5 or day 6.
  Treatment Weeks 13-18: Mifamurtide 2mg/m2, IV infusion, twice/week. Treatment Weeks 19-42: Mifamurtide 2mg/m2, IV infusion, once/week.
  Mifamurtide
  Ifosfamide
- C. Ifosfamide + Mifamurtide: Patients receive mifamurtide combined with ifosfamide initially.
  Treatment Weeks 1-6:
  Day 1 of 21: Ifosfamide 12-15g/m2 IV infusion infused over 4-5 days once every 21 days for two cycles (3 weeks=1 cycle).
  Plus Mifamurtide 2 mg/m2, IV infusion, twice per week, with each infusion given at least 3 days apart, for 6 weeks.
  Ifosfamide infusion must be started 24 hours prior to mifamurtide. Mifamurtide should be given on day 2 and either day 5 or day 6.
  Treatment Weeks 7-12 (post 2nd biopsy/resection):
  Day 1 of 21: Ifosfamide 12-15g/m2 IV infusion infused over 4-5 days once every 21 days for two cycles (3 weeks = 1 cycle).
  Plus Mifamurtide 2mg/m2, IV infusion, twice per week, with each infusion given at least 3 days apart, for 6 weeks. Ifosfamide infusion must be started 24 hours prior to mifamurtide. Mifamurtide should be given on day 2 and either day 5 or day 6.
  Treatment Weeks 13-36: Mifamurtide 2mg/m2, IV infusion, once/week.
  Mifamurtide
  Ifosfamide
Period: Overall Study
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Started | 3 | 2 | 3
Received Allocated Intervention | 1 | 2 | 3
Completed | 0 | 0 | 0
Not Completed | 3 | 2 | 3
Not completed — Disease progression | 2 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide | Total
Number analyzed (Participants) | 3 | 2 | 3 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [20 to 22] | 23 [20 to 25] | 57 [41 to 59] | 25 [20 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 3 | 2 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 0 | 0 | 1 | 1
  Norway | 1 | 0 | 1 | 2
  United Kingdom | 1 | 2 | 1 | 4
  Italy | 1 | 0 | 0 | 1
WHO Performance Status [Count of Participants; unit: Participants] — WHO performance status classification
  The WHO performance status classification categorises patients as:
  0. able to carry out all normal activity without restriction
  1. restricted in strenuous activity but ambulatory and able to carry out light work
  2. ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. symptomatic and in a chair or in bed for greater than 50% of the day but not bedridden
  4. completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0 | 3 | 1 | 2 | 6
    1 | 0 | 1 | 1 | 2
Histology/Cytological type [Count of Participants; unit: Participants] — International classification of diseases for oncology. ICD-O-3 online
  Participants
    Chondroblastic OS - 9181/3 | 1 | 0 | 0 | 1
    Osteoblastic OS - 9180/3 | 1 | 0 | 1 | 2
    Osteosarcoma NOS - 9180/3 | 1 | 2 | 2 | 5
Primary Site [Count of Participants; unit: Participants]
  Axial | 1 | 1 | 1 | 3
  Limb | 2 | 1 | 2 | 5
Disease stage at screening - Metastatic [Count of Participants; unit: Participants] | 3 | 2 | 3 | 8
Tumour size at baseline (sum of longest diameters) (mm) [Median (Inter-Quartile Range); unit: mm] | 84 [83 to 84] | 37 [33 to 42] | 99 [78 to 174] | 82 [81 to 92]
Prior chemotherapy [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1 | 2
  No | 2 | 2 | 2 | 6
Prior radiotherapy [Count of Participants; unit: Participants]
  Yes | 3 | 2 | 3 | 8
  No | 0 | 0 | 0 | 0
Prior surgery [Count of Participants; unit: Participants]
  Yes | 3 | 2 | 3 | 8
  No | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Biological Response Data Based on Pharmacodynamic Endpoints on Tumour Biopsy Material
Description: Biological response data based on pharmacodynamic endpoints on tumour biopsy material including macrophage infiltration and innate immune activation.
Time Frame: Change from Baseline to after 6 weeks of treatment
Population: Insufficient number of participants for events for both primary and secondary objectives. The study stopped prematurely because of poor recruitment, meaning that no complete statistical analysis was possible as there were insufficient events and data were not collected.
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Radiological Response Defined as Complete or Partial Response and Assessed Using RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) assessed by CT or MRI:
  Complete Response (CR): Disappearance of all target and non-target lesions Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions, AND no evidence of progression in non-target lesions, AND no new lesions Stable Disease (SD): sum of longest diameter of target lesions between PR and PD values, AND no evidence of progression in non-target lesions, AND no new lesions Progressive Disease (PD): >20% increase in the sum of the longest diameter of target lesions, OR evidence of progression in non-target lesions, OR evidence of new lesions
Time Frame: Change from Baseline to after 6 weeks of treatment
Population: All patients are included since this is an intention to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 3 | 2 | 3
Participants
  Stable Disease (SD) | 0 | 1 | 1
  Progressive Disease (PD) | 0 | 0 | 1
  Patient did not reach endpoint | 1 | 1 | 1
  Patient progressed prior to time point | 2 | 0 | 0

3. Secondary Outcome: Objective Radiological Response Based on RECIST v1.1
Description: as for outcome 2
Time Frame: Change from Baseline to after 12, 18, 24 & 36 weeks and end of treatment visit
Population: The end of treatment visit was completed by patients who were deemed to progress or withdrew from trial treatment at a time that a scheduled scan was not due to be taken. This end of treatment visit was used to confirm radiological progression.
Measure: Count of Participants; unit: Participants
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 3 | 2 | 3
Participants
  Week 12: Stable Disease (SD) | 0 | 1 | 1
  Week 12: Progressive Disease (PD) | 0 | 0 | 0
  Week 12: Patient did not reach endpoint | 3 | 1 | 2
  Week 18: Stable Disease (SD) | 0 | 1 | 0
  Week 18: Progressive Disease (PD) | 0 | 0 | 1
  Week 18: Patient did not reach endpoint | 3 | 1 | 2
  Week 24: Stable Disease (SD) | 0 | 1 | 0
  Week 24: Progressive Disease (PD) | 0 | 0 | 0
  Week 24: Patient did not reach endpoint | 3 | 1 | 3
  Week 36: Stable Disease (SD) | 0 | 0 | 0
  Week 36: Progressive Disease (PD) | 0 | 1 | 0
  Week 36: Patient did not reach endpoint | 3 | 1 | 3
  End of Treatment visit (prior to week 6): number analyzed (Participants) | 2 | 0 | 0
  End of Treatment visit (prior to week 6): Stable Disease (SD) | 0 | 0 | 0
  End of Treatment visit (prior to week 6): Progressive Disease (PD) | 2 | 0 | 0
  End of Treatment visit (prior to week 6): Patient did not reach endpoint | 0 | 0 | 0

4. Secondary Outcome: Number of Patients Experiencing a Grade 3 or More Severe Adverse Event (Graded According to CTCAE Criteria v4.0)
Description: Toxicity measured and graded according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
  Grade refers to the severity of the adverse event. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 Severe; medically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation indicated; disabling or limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Up to 42 weeks
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 3 | 2 | 3
Participants | 1 | 2 | 2

5. Secondary Outcome: Number of Patients Experiencing a Laboratory Abnormality (Grade 3-4)
Description: A laboratory abnormality is defined as an adverse event of grade 3 or 4 identified by a laboratory test of participant blood samples.
  Adverse events were graded according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
Time Frame: Up to 42 weeks
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 3 | 2 | 3
Participants | 0 | 0 | 0

6. Secondary Outcome: Disease Specific Overall Survival
Description: Median time from death attributed to the disease. Censored at last known time alive or death from other causes.
Time Frame: Up to 42 weeks
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 3 | 2 | 3
months | 0.7 [0.2 to NA] — Undefined upper confidence interval (insufficient number of participants with events). | 9.2 [9.2 to NA] — Undefined upper confidence interval (insufficient number of participants with events). | 2.8 [1.5 to NA] — Undefined upper confidence interval (insufficient number of participants with events).

7. Secondary Outcome: Progression Free Survival
Description: Time from randomisation for deemed non-resectable groups, or time from registration for deemed resectable group to first event, where an event is Progressive Disease as (defined by RECIST criterion v1.1) or death due to any cause. Patients who have not had an event will be censored at their last follow-up date. Patients lost to follow-up without an event will be censored at the date of their last consultation.
  Progressive disease according to RECIST v1.1 is defined as a >=20% increase in the sum of long diameters of target lesions, OR progression of non-target lesions, OR evidence of new lesions.
Time Frame: Up to 42 weeks
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 3 | 2 | 3
months | NA [NA to NA] — No events were observed, median is undefined. | NA [NA to NA] — No events were observed, median is undefined. | 7.0 [4.6 to NA] — Undefined upper confidence interval (insufficient number of participants with events).

8. Secondary Outcome: Biological Response (Systemic Levels of Mifamurtide Activated Cytokines).
Description: Biological response based on systemic levels of mifamurtide activated cytokines.
Time Frame: During screening, and weeks 1, 4, 6 and 7. Then every 3 weeks during treatment.
Population: as for outcome 1
Groups:
- A. Mifamurtide Only: Treatment Weeks 1-6 (post 1st biopsy/resection):
  Mifamurtide 2mg/m2, IV infusion, twice/week, with each infusion given at least 3 days apart, for 6 weeks.
  Treatment Weeks 7-12 (post 2nd biopsy/resection):
  Mifamurtide 2mg/m2, IV infusion, twice/week, with each infusion given at least 3 days apart, for 6 weeks.
  Treatment Weeks 13-36:
  Mifamurtide 2mg/m2, IV infusion, once/week.
  Mifamurtide
- B. Ifosfamide (Followed by Mifamurtide): Treatment Weeks 1-6: Day 1 of 21: Ifosfamide 12-15g/m2 IV infused over 4-5 days as per local practice. Repeated every 21 days for 2 cycles (3 weeks=1 cycle).
  Treatment Weeks 7-12 (post 2nd biopsy/resection): Day 1 of 21: Ifosfamide 12-15g/m2 IV infused over 4-5 days once every 21 days for two cycles (3 weeks=1 cycle). Ifosfamide administered as per local practice, including concurrent dosing with mesna. Plus mifamurtide 2mg/m2, IV infusion, twice/week. Ifosfamide infusion started 24 hours prior to mifamurtide. Mifamurtide given on day 2 and either day 5 or day 6.
  Treatment Weeks 13-18: Mifamurtide 2mg/m2, IV infusion, twice/week. Treatment Weeks 19-42: Mifamurtide 2mg/m2, IV infusion, once/week.
  Mifamurtide
  Ifosfamide
- C. Ifosfamide + Mifamurtide: Treatment Weeks 1-6:
  Day 1 of 21: Ifosfamide 12-15g/m2 IV infusion over 4-5 days once every 21 days for two cycles (3 weeks=1 cycle).
  Plus Mifamurtide 2mg/m2, IV infusion, twice per week, each given at least 3 days apart, for 6 weeks.
  Ifosfamide infusion started 24 hours prior to mifamurtide. Mifamurtide given on day 2 and either day 5 or day 6.
  Treatment Weeks 7-12 (post 2nd biopsy/resection):
  Day 1 of 21: Ifosfamide 12-15g/m2 IV infusion over 4-5 days once every 21 days for two cycles (3 weeks = 1 cycle).
  Plus Mifamurtide 2mg/m2, IV infusion, twice per week, given at least 3 days apart, for 6 weeks. Ifosfamide infusion started 24 hours prior to mifamurtide. Mifamurtide given on day 2 and either day 5 or day 6.
  Treatment Weeks 13-36: Mifamurtide 2mg/m2, IV infusion, once/week.
  Mifamurtide
  Ifosfamide
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from registration until the end of treatment (42 weeks) or the withdrawal of treatment.
Description: An abnormal laboratory value will not be assessed as an AE unless that value leads to discontinuation or delay in treatment, dose modification, therapeutic intervention, or is considered by the investigator to be a clinically significant change from baseline.
Arm/Group | A. Mifamurtide Only | B. Ifosfamide (Followed by Mifamurtide) | C. Ifosfamide + Mifamurtide
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/2 | 2/3
Other Adverse Events (participants affected / at risk) | 1/3 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A. Mifamurtide Only (N=3) | B. Ifosfamide (Followed by Mifamurtide) (N=2) | C. Ifosfamide + Mifamurtide (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A. Mifamurtide Only (N=3) | B. Ifosfamide (Followed by Mifamurtide) (N=2) | C. Ifosfamide + Mifamurtide (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1
Fever (General disorders) | 1 | 0 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0
Shivering (General disorders) | 0 | 0 | 1
Central line infection (Infections and infestations) | 0 | 1 | 0
Infected toe (Infections and infestations) | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Taste altered (Nervous system disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. This was due to a poor recruitment speed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes